CLINICAL TRIAL: NCT06247150
Title: Tissue Immune Landscape of Graft Versus Host Disease After Allogeneic Stem Cell Transplantation (TIL-GVHD)
Acronym: TIL-GVHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHUBX 2021/15
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: Chronic GVHD; Biopsy; TFH; Tertiary lymphoid structures
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Tertiary Lymphoid Structures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with cGVHD (Other)
  Interventions: Biological: Additional blood sample; Biological: cGVHD target tissue biopsy
- Patients without cGVHD (Other)
  Interventions: Biological: Additional blood sample

INTERVENTIONS:
Biological: Additional blood sample — The procedure will consist of an additional blood sample for 3 ETDA tubes collection (NGS analysis) and citrate tube collection (NETose analysis)
Biological: cGVHD target tissue biopsy — For chronic GVH patients only, cGVHD target tissue biopsy
  Arms: Patients with cGVHD

SUMMARY:
Graft versus Host Disease (GVHD) is frequent after allogeneic stem cell transplantation (alloSCT). GVHD occurs following 2 patterns : acute GVHD (aGVHD) or chronic GVHD (cGVHD). The latter occurs in nearly 50% of patients and its pathogenesis remains poorly understood. Previous translational studies have delineated biological immune dysregulation involved in cGVHD and facilitated the development of new drug and therapeutic strategies. New aspects of T and B cells collaboration in the context of cGVHD using blood description of a key player called TFH, classicaly involved in germinal center reaction, were previously uncovered (Forcade et al, Blood 2016). Previous studies in the context of auto-immune inflammation (lupus nephritis) or organ transplant rejection, suggested that target tissue could contain accessory lymphoid structures (TLS). The description of such structures in cGVHD target tissue would give the opportunity to directly analyze immune key player involved the pathogenesis of cGVHD.

DETAILED DESCRIPTION:
Context :

Chronic Graft versus Host Disease (cGVHD) represents the main cause of morbidity and mortality in patients undergoing hematopoietic stem cell transplantation (alloSCT), occurring in 30 and 60%. Translational studies showed that different alloreactive T cell subsets were involved and associated with cGVHD, and regulatory subsets were deficient. Several homeostatic abnormalities of B cell subsets were also shown, which, in the context of high BAFF level, contributed to autoreactive B cell clone emergence.

In alloSCT patients, we observed (Forcade et al, Blood 2016) in the blood, a T cell subset called TFH, with B cell help capacity, similar to germinal center reaction. During cGVHD, blood TFH were highly activated, skewed toward a Th1/Th17 profile, and presented enhanced capacity to provide " help " to B cells, promoting auto-/allo-antibody production in the context of cGVHD. This was associated with increased level of CXCL13 in such patients, suggesting homing of this subset to lymphoid tissues.

Liarski et al (Sci Trans Med 2014) showed that TFH were observed in inflamed tissue sample from patients with lupus, and demonstrated close interaction with B cells, mimicking germinal center structures, such as tertiary lymphoid organs.

Preliminary data, on cGVHD tissue target, showed a CD4+ T cell infiltrate, of which some expressed CXCR5, ICOS, PD1 in single staining.

Hypothesis : cGVHD target tissue contains tertiary lymphoid structures.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 yo ;
* Having undergone an allogeneic stem cell tranplant ;
* 2 groups of patients will be eligible
* showing evidence of primary cGVHD or occuring after Donor Lymphocyte Infusion

  * in the case of first occurrence of cGVHD, in the absence of any new systemic therapy ;
  * in the case of recurrent cGVHD, steroid dose has to be below 15mg/day of Prednisone ;
* Having read, understood and signed an informed consent of the study;
* With social security affiliation;

Exclusion Criteria:

* Patient below 18 yo or unable to give consent ;
* Systemic therapy using steroids over 15mg/d of Prednisone ; and/or the use of other systemic agent introduced in the last month ;
* Haemorrhagic risk of biopsy anticipated ;
* Absence of patient agreement for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
To describe immune landscape in chronic GVHDtarget tissuesubsets, especially TFH, within cGVHD tissue target, using flow cytometry and histology | At inclusion visit
  Flow cytometry and multiplex tissue imaging. GVHD evaluation using NIH score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Service d'Hématologie Clinique et Thérapie Cellulaire, Pessac, France

IPD SHARING:
Plan to Share IPD: No